CLINICAL TRIAL: NCT01057433
Title: Drug-Drug Interaction Study to Assess the Effects of Steady-State Lopinavir/Ritonavir on Pitavastatin in Healthy Adult Volunteers
Brief Title: Drug-Drug Interaction of Lopinavir/Ritonavir on Pitavastatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NK-104-4.02US
Record Dates: First submitted 2010-01-25; First posted 2010-01-27 (Estimated); Results first posted 2012-08-13 (Estimated); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — pitavastatin; Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pitavastatin (Experimental): Healthy adult subjects
  Interventions: Drug: Pitavastatin (NK-104); Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Pitavastatin (NK-104) — pitavastatin (NK-104) 4 mg once daily (QD)
  Other Names: Livalo
Drug: Lopinavir/ritonavir — lopinavir/ritonavir 800 mg/200 mg
  Other Names: Kaletra

SUMMARY:
This is a Phase 4, single center, open label, fixed-sequence, 2-way drug-drug interaction study.

DETAILED DESCRIPTION:
This is a Phase 4, single center, open label, fixed-sequence, 2-way drug-drug interaction study.

Each subject will qualify for entry into the study not more than 30 days prior to admission into the clinical unit. Subjects will check into the clinical unit on Day -1 for baseline assessments. There will be one treatment period, with each subject receiving a once daily dose of pitavastatin 4 mg on Days 1 through 5 and Days 20 through 24 and a twice daily dose of lopinavir/ritonavir 400 mg/100 mg (two 200 mg/50 mg tablets per dose) on Days 9 through 24. Pitavastatin will be administered under fasting conditions in the morning and lopinavir/ritonavir will be administered under fasting conditions in the morning and evening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteer aged 18 to 45 years, inclusive.
* Subject has a body mass index of 18 to 30 kg/m2, inclusive.
* Subject has normal hematology, serum chemistry, and urinalysis test results
* Subject is able and willing to abstain from alcohol, grapefruit, caffeine, or caffeine containing products for 4 days before Day 1 until after completion of this study.
* Subject is a nonsmoker or has quit smoking at least 6 months before the first dose of study drug.

Exclusion Criteria:

* Subject has had any surgery of the gastrointestinal tract likely to affect drug absorption, distribution, metabolism, or excretion.
* Subject has had a previous allergy or intolerance to treatment with pitavastatin or lopinavir/ritonavir.
* Subject has a history of drug or alcohol abuse.
* Subject has had a clinically significant illness within 4 weeks before the first dose of study drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Morgan, MD, FACS, Study Director — Kowa Research Institute, Inc.
Locations (1):
- Austin, Texas, United States

REFERENCES:
- [Derived] Morgan RE, Campbell SE, Suehira K, Sponseller CA, Yu CY, Medlock MM. Effects of steady-state lopinavir/ritonavir on the pharmacokinetics of pitavastatin in healthy adult volunteers. J Acquir Immune Defic Syndr. 2012 Jun 1;60(2):158-64. doi: 10.1097/QAI.0b013e318251addb. PMID 22627182

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 24
Completed | 23
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to Tau (AUC 0-τ)
Description: Area under the curve from start to elimination.
Time Frame: 0, 1, 2, 3, 4, 5, 6, 8, and 12 hours after dosing on days 19 and 24
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | All Subjects
Number analyzed (Participants) | 23
ng•h/mL | 113.92 (53.80)

ADVERSE EVENTS:
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 18/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Subjects (N=24)
Diarrhea (Gastrointestinal disorders) | 13
Abdominal pain (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 8
Anal hemorrhage (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3
Rash macular (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
May not publish.